CLINICAL TRIAL: NCT02800369
Title: Safety Study of Zinc Finger Nucleases ZFN-602 and ZFN-758 in HPV-infected Subjects
Brief Title: Study of Molecular-targeted Therapy Using Zinc Finger Nuclease in Cervical Precancerous Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Head of Cancer Biology center, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016ZFN-V02
Record Dates: First submitted 2016-06-01; First posted 2016-06-15 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Human Papillomavirus-Related Malignant Neoplasm
Keywords: Human papillomavirus; cervical intraepithelial neoplasia; zinc finger nuclease
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZFN-603 and ZFN-758 (Experimental): Subjects will receive suppository with ZFN-603 or ZFN-758
  Interventions: Biological: ZFN-603 and ZFN-758

INTERVENTIONS:
Biological: ZFN-603 and ZFN-758 — Each suppository contain 500 µg of ZFN-603 or ZFN-758

SUMMARY:
This research study is being carried out to study a new way to possibly treat human cervical intraepithelial neoplasia (CIN) without invasion.

Persistent infection with specific types of human papillomavirus (HPV, most frequently types 16 and 18) may lead to precancerous lesions(CIN). If untreated, these lesions may progress to cervical cancer within many years. In the infected cells, HPV expresses the oncoproteins E6 and E7, both of which play key roles in maintaining viral infection and promoting carcinogenesis. Previous studies has demonstrated that E7 alone, but not E6, is sufficient to immortalize human keratinocytes in vitro and induce high-grade cervical dysplasia in a transgenic mouse model. These data indicated that E7 may dominate the malignant progress in HPV-infected cells.

The agents zinc finger nucleases (ZFNs), called ZFN-603 and ZFN-758, which can cleave the HPV16 and HPV18 E7 oncogene specifically. ZFN-mediated disruption of HPV16 and HPV18 E7 DNA directly decreased the expression of E7, induced type-specific apoptosis in HPV16- and HPV18-positive cells, and inhibited cell growth.

The purpose of this study is to determine whether ZFN-603 and ZFN-758 are effective in the treatment of HPV16- and HPV18-positive cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
Laboratory studies have shown that ZFN-603 and ZFN-758 could induce significant cleavage of E7 DNA in HPV16- and HPV18-positive cells. The disruption to viral DNA directly led to downregulation of E7 expression and restoration of the tumor suppressor genes retinoblastoma 1 (RB1), resulting in apoptosis and growth inhibition of ZFN-treated HPV16- and HPV18- positive cell lines. On the basis of these laboratory results, there is the potential that this may work in humans infected with high-risk HPV (especially HPV16 and HPV18) and block the progression of CIN The new treatment to be studied will involve transfecting ZFNs into HPV-infected cervical epithelials. Cells modified by ZFN-603 and ZFN-758 will lose the ability of immortalization and progress to apoptosis.

Researchers hope that these agents will be able to block the malignant progression of CIN and reduce the incidence of cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Documented HPV16 or HPV18 infection.
* Married and fertile, no fertility requirements.
* Without administration of hormone in the last six months
* Subjects must be meet the ethical requirements and have signed informed consent

Exclusion Criteria:

* Pregnancy and breast feeding
* Any bacterial vaginitis
* Any Fungal vaginitis
* Any sexually transmitted diseases
* Active drug or alcohol abuse
* Any HPV medications within the past 12 weeks
* Allergy to active or non active ingredients in the study of drugs
* Cardiac insufficiency
* Liver and renal insufficiency
* Hypertension and severe complications
* Serious illness in past 30 days
* Currently participating in another clinical trail or any prior gene therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12-10 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-07-10 (Estimated)

PRIMARY OUTCOMES:
Safety - Treatment related adverse events of ZFN-603 in HPV16-positive subjects, related adverse events of ZFN-758 in HPV18-positive subjects | 6 months
  Number of participants who report adverse events as a measure of safety

SECONDARY OUTCOMES:
Evaluate persistence of HPV16 and HPV18 as measured by HPV DNA | 6 months
  Reduce the virus titers after using ZFN-603 and ZFN-758
Change in the number of dysplastic cells as mearsured by ThinPrep Pap Test | 6 months
  From high-grade squamous intraepithelial lesion (HSIL) to Low-grade Squamous Intraepithelial Lesion (LSIL), or from LSIL to negative.
Number of participants with Regain health or without progress | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, M.D., Study Director — Huazhong University of Science and Technology; Wencheng Ding, M.D., Principal Investigator — Huazhong University of Science and Technology; Da Zhu, M.D., Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ding W, Hu Z, Zhu D, Jiang X, Yu L, Wang X, Zhang C, Wang L, Ji T, Li K, He D, Xia X, Liu D, Zhou J, Ma D, Wang H. Zinc finger nucleases targeting the human papillomavirus E7 oncogene induce E7 disruption and a transformed phenotype in HPV16/18-positive cervical cancer cells. Clin Cancer Res. 2014 Dec 15;20(24):6495-503. doi: 10.1158/1078-0432.CCR-14-0250. Epub 2014 Oct 21. PMID 25336692